CLINICAL TRIAL: NCT03081572
Title: Differences in Platelet Function in Patients on Abacavir Versus Tenofovir Based Antiretroviral Regimens
Brief Title: Platelet Function on Abacavir and Tenofovir
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 5P30A1028697
Record Dates: First submitted 2017-03-01; First posted 2017-03-16 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Cardiovascular Diseases; Platelet Aggregation, Spontaneous; HIV/AIDS
MeSH Terms: conditions — Cardiovascular Diseases; Platelet Aggregation, Spontaneous; Acquired Immunodeficiency Syndrome | interventions — Platelet Aggregation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Abacavir Group: HIV positive individuals currently taking an abacavir based regimen
  Interventions: Diagnostic Test: Platelet aggregation
- Tenofovir Group: HIV positive individuals currently taking a tenofovir based regime
  Interventions: Diagnostic Test: Platelet aggregation

INTERVENTIONS:
Diagnostic Test: Platelet aggregation — Platelet aggregation

SUMMARY:
This is a small observational study aimed at observing differences in platelet function in HIV patients on abacavir versus tenofovir based anti-HIV drugs. There is some correlation between platelet activation and cardiovascular disease- this study will act as a pilot to see if platelet activation among abacavir users may explain the correlation between abacavir and cardiovascular disease in HIV positive patients.

This study will enroll 44 participants total; 22 on abacavir-based treatment, 22 on tenofovir-based treatment. There is only one study visit which includes a blood draw, physical assessment, and review of medical history.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive
* Stable antiretroviral regimen for > 3months containing either abacavir or tenofovir
* Suppressed HIV viral load

Exclusion Criteria:

* Current cigarette smoking
* Pre-existing platelet disorder
* current or recent (last 6 months) antiplatelet therapy
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV positive non smokers who are on a stable antiretroviral regimen containing either abacavir or tenofovir
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-04-30 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-02-15 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation | At screening visit
  Degree of platelet aggregation in response to adenosine diphosphate

SECONDARY OUTCOMES:
Plasma Markers of coagulation | At screening visit
  sGPVI
Plasma Markers of Coagulation | At screening visit
  sPSelectin
Plasma markers of endothelial function | At screening visit
  sICAM

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical AIDS Research and Education Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data